CLINICAL TRIAL: NCT07290270
Title: Real-world Use of Lutetium (177Lu) Vipivotide Tetraxetan Injection in Metastatic Prostate Cancer: an Observational, Multicenter, Prospective Cohort Study in China (PSMAreal CN)
Brief Title: Real-world Use of Lutetium (177Lu) Vipivotide Tetraxetan in China(PSMAreal CN)
Acronym: PSMAreal
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA617A1CN01
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer; Metastatic Hormone-Sensitive Prostate Cancer; Lutetium (177Lu) vipivotide tetraxetan Injection; Non-interventional Study; China
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Patients diagnosed with Metastatic Castration-Resistant Prostate Cancer (mCRPC) previously treated with at least one ARPI with or without taxane regimens.
- Cohort 2: Patients diagnosed with Metastatic Hormone-Sensitive Prostate Cancer (mHSPC).

SUMMARY:
This non-interventional, observational, multicenter, prospective cohort study is designed to investigate the treatment patterns of mPC patients treated with lutetium (177Lu) vipivotide tetraxetan, as well as their clinical outcomes, real-world characteristics, and quality of life during the treatment period and up to one year after treatment completion.

DETAILED DESCRIPTION:
The study population will be divided into two cohorts, enrolling patients with mCRPC and mHSPC, respectively. Patients planned to receive lutetium (177Lu) vipivotide tetraxetan treatment according to treating physician's assessment will be enrolled in the study upon signing an informed consent form. Patients must meet all inclusion criteria defined in the protocol and not meet any exclusion criteria. The patients' medical history, prostate cancer disease characteristics, demographics, and baseline data will be collected through medical records and examination reports. Treatment patterns, treatment outcomes, and HRQoL data will be collected during study follow-up visits through patient records, examination reports, and self-reported data. This study does not have a control group; instead, a self-control method will be used, with the patients' baseline data before the start of treatment serving as the control for efficacy, safety, and HRQoL assessments. The index date for this study is defined as the date of the first administration of lutetium (177Lu) vipivotide tetraxetan

ELIGIBILITY:
Inclusion Criteria:

Adult male patients diagnosed with mCRPC or mHSPC Initiating lutetium (177Lu) vipivotide tetraxetan treatment by treating physician as per local label. After treatment decision enrollment is allowed before date of cycle 1 or within 2 weeks after the date of cycle 1 Written ICF must be obtained prior to any data collection Participants must have adequate organ function following Society of Nuclear Medicine and Molecular Imaging (SNMMI) consensus (Hope et al., 2023)

Exclusion Criteria:

Simultaneous participation in any investigational trial or simultaneous participation in another Novartis-sponsored non-interventional study with lutetium (177Lu) vipivotide tetraxetan during the study period

Other protocol-defined inclusion / exclusion criteria may apply

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients
Study Population: The study population will be recruited from approximately 25 research centers in China
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
prostate-specific antigen (PSA) 50 response rate | from 1 month before the index date through to 1 year after the end-of-treatment (EOT) visit
  Defined as the proportion of patients with a confirmed decrease in PSA levels by ≥50% from baseline
prostate-specific antigen (PSA) 90 response rate | from 1 month before the index date through to 1 year after the end-of-treatment (EOT) visit
  Defined as the proportion of patients with confirmed decreases in PSA level by ≥90% from baseline

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the first occurrence of PSA progression or radiographic progression according to the Prostate Cancer Working Group 3 criteria, clinical progression assessed by the investigator, or death due to any cause (whichever occurs first)
Radiographic progression-free survival (rPFS) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the first occurrence of radiographic progression according to the PCWG3 criteria or death due to any cause (whichever occurs first)
Clinical PFS | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the first occurrence of clinical progression assessed by the investigator or death due to any cause (whichever occurs first). Clinical progression is determined by the investigator and may be based on the following criteria: 1) Significant increase in tumor pain requiring initiation of another systemic anti-cancer treatment regimen; 2) The need to immediately start new anti-cancer treatment, surgery, or radiotherapy intervention due to complications caused by tumor progression, even in the absence of radiographic progression; 3) Deterioration of Eastern Cooperative Oncology Group (ECOG) performance status to ≥ 3, and the investigator determines that the deterioration indicates clinical progression
Time to PSA progression | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the first occurrence of PSA progression or death due to any cause. According to the PCWG3 criteria, PSA progression is defined as follows:
  1. For patients whose PSA has declined from baseline: PSA increased by ≥25% compared with the lowest value and the absolute value was ≥2 ng/mL, and was re-evaluated and confirmed after ≥3 weeks.
  2. For patients whose PSA has not declined from baseline: After at least 12 weeks of treatment with the study drug, the PSA level increased by ≥25% from the baseline and the absolute value was ≥2 ng/mL
Second Progression-Free Survival (PFS2) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the initiation of the first subsequent systemic anti-tumor therapy following the end of treatment with lutetium (177Lu) vipivotide tetraxetan to the first occurrence of radiographic progression or PSA progression according to the PCWG3 criteria, clinical progression as assessed by the investigator, or death due to any cause (whichever occurs first)
OS | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to death due to any cause
Time to a first symptomatic skeletal event (SSE) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the first occurrence of an SSE. SSEs include the use of external beam radiation therapy to prevent or palliate skeletal symptoms, the occurrence of a new symptomatic pathological fracture (vertebral or non-vertebral), the occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention (whichever occurs first)
Time to first subsequent therapy | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the start date of the first subsequent therapy for prostate cancer. Subsequent therapy refers to systemic anti-tumor treatment initiated after the patient discontinues lutetium (177Lu) vipivotide tetraxetan treatment
Disease control rate (DCR) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the proportion of patients with complete response (CR) / partial response (PR), and stable disease (SD) as the best response in soft tissue lesion evaluation
Objective response rate (ORR) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the proportion of patients with CR and PR as the best response in soft tissue lesion evaluation assessed referring to the evaluation criteria
Time to response (TTR) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the first documentation of CR or PR for soft tissue lesions referring to the evaluation criteria
Duration of response (DoR) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the first documentation of objective response (CR or PR) to the first occurrence of disease progression (radiographic, clinical, or PSA progression) or death due to any cause (whichever occurs first)
Time to soft tissue progression (TTSTP) | Data collection for radiographic assessment outcomes: from 3 months before the index date to 1 year after the EOT visit / Data collection for non-radiographic assessment outcomes: from 1 month before the index date to 1 year after the EOT visit
  Defined as the time from the index date to the occurrence of soft tissue progression referring to the evaluation criteria or death due to any cause (whichever occurs first)
Number of participants by treatment dose and cycles of lutetium (177Lu) vipivotide tetraxetan | Data collection of previous treatments for prostate cancer: from the time of prostate cancer diagnosis to the index date / Data collection of subsequent treatments for prostate cancer: from the index date to 1 year after the EOT visit
  Number of participants by treatment dose and cycles of lutetium (177Lu) vipivotide tetraxetan
Number of participants by treatment sequences for prostate cancer | Data collection of previous treatments for prostate cancer: from the time of prostate cancer diagnosis to the index date / Data collection of subsequent treatments for prostate cancer: from the index date to 1 year after the EOT visit
  Prior treatment lines and subsequent treatments (including: ARPI, ADT, chemotherapy, radical prostatectomy, radiological treatment etc.)
Patient demographics and baseline characteristics | From 1 month before the index date to the index date
Prostate cancer disease characteristics: Number of patients with Previous prostate cancer history | Baseline
Prostate cancer disease characteristics: Gleason score | From 1 month before the index date to the index date
  Typical Gleason Scores range from 6-10. The higher the Gleason Score, the more likely that the cancer will grow and spread quickly.
Prostate cancer disease characteristics: Number of patients by metastasis status | From 1 month before the index date to the index date
Prostate cancer disease characteristics: Number of patients by prostate cancer-related genetic mutation status | From 1 month before the index date to the index date
Prostate cancer disease characteristics: Baseline prostate-specific antigen (PSA) level | Baseline
Prostate cancer disease characteristics: prostate-specific antigen (PSA) doubling time | From 1 month before the index date to the index date
Prostate cancer disease characteristics: Prostate-Specific Membrane Antigen (PSMA) diagnostic drug usage | From 1 month before the index date to the index date
Prostate cancer disease characteristics: Baseline PET-CT results | Baseline
Prostate cancer disease characteristics: Baseline testosterone level | Baseline
Prostate cancer disease characteristics: Baseline Eastern Cooperative Oncology Group (ECOG) performance status | Baseline
  ECOG performance status is measured on a 6 point grade scale.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
Prostate cancer disease characteristics: Number of patients with family history of prostate cancer | Baseline
Prostate cancer disease characteristics: Number of patients with carcinoembryonic Antigen (CEA) | From 1 month before the index date to the index date
Adverse events | From the index date to 1 year after the EOT visit
FACT-P score | From 1 month before the index date to 1 year after the EOT visit
  The FACT-P was developed to measure the health-related quality of life (HRQOL) in patients diagnosed with prostate cancer. It extends the general FACT-G scale, which assesses cancer patients' overall quality of life, by adding specific items related to prostate cancer therapy. The FACT-P consists of two main sections:
  1. FACT-G: A general section that covers four domains: Physical Well-Being (PWB)，Social/Family Well-Being (SWB)，Emotional Well-Being (EWB)，Functional Well-Being (FWB)
  2. Prostate Cancer Specific Section: Focuses on issues unique to prostate cancer patients, such as urinary symptoms, sexual health, and the side effects of treatment.
  The scoring system for the FACT-P uses a 5-point Likert scale (from 0 to 4，from good to bad). Scores are calculated across different domains and subscales, and the total score is calculated by summing the scores across all domains, providing a range of 0 to 156. A high FACT-P score indicates a worse outcome.
BPI-SF score | From 1 month before the index date to 1 year after the EOT visit
  Brief Pain Inventory-Short Form (BPI-SF). The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning. BPI assessment areas including severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
EQ-5D-5L questionnaire score | From 1 month before the index date to 1 year after the EOT visit
  EuroQol 5-Dimension 5-Level (EQ-5D-5L). The 5-level EQ-5D version (EQ-5D-5L) descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
FACT-RNT score | From 1 month before the index date to 1 year after the EOT visit
  Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT). The FACT-RNT was designed for use and future adaptation with a broad variety of RNT agents with different molecular targeting mechanisms and radioisotopes. The FACT-RNT, a 15-item measure of symptoms/toxicities with higher total scores(range:0-60) indicating less symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pjharmaceuticals, Study Director — Novartis Pjharmaceuticals

IPD SHARING:
Plan to Share IPD: No